CLINICAL TRIAL: NCT02895568
Title: Prevalence Survey of Plasmodium Falciparum Antimalarial Drug Resistance Markers in Komé, Doba, Republic of Chad
Brief Title: Prevalence Survey of Plasmodium Falciparum Antimalarial Drug Resistance Markers
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Worldwide Antimalarial Resistance Network (Network); Mahidol University (Other)
Responsible Party: Sponsor
Other Study IDs: WWARN1603
Record Dates: First submitted 2016-08-22; First posted 2016-09-09 (Estimated); Last update posted 2022-04-07 (Actual); Status verified 2018-11

CONDITIONS: Plasmodium Falciparum
Keywords: Antimalarial drug; Resistance; Republic of Chard
MeSH Terms: conditions — Malaria, Falciparum

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — A dried blood spot sample for study analyses will be collected at the time of blood collection for malaria diagnostic testing.
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is to measure prevalence of established and candidate molecular markers of drug resistant malaria at Komé, Doba, Republic of Chad.

DETAILED DESCRIPTION:
This is a cross-sectional, observational study using dried blood samples collected from P. falciparum-infected individuals at the time of malaria diagnosis to measure the prevalence of known and candidate molecular markers of resistance to artemisinin and non-artemisinin ACT partner drugs. A maximum of 200 participants will be enrolled at each participating site per year. Study duration is 2 years. Therefore total participant is up to 400.

Prospective participants will have blood collected for dried blood spot (DBS) study sample after providing informed consent. Individuals with confirmed P. falciparum infection will have DBS samples included for molecular analyses for known and candidate molecular markers of antimalarial drug resistance.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the inclusion criteria to participate in the study.

* Patients (6 months - 75 years) with confirmed uncomplicated P. falciparum infection
* Written informed consent obtained

Exclusion Criteria:

* Patients presenting signs of severe malaria will be excluded from the survey to prevent any delay in the management of the patient.

Ages: 6 Months to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study participants will be the patients presenting at study clinics with signs and symptoms of malaria (including but not limited to headache, body aches, fever, chills, and weakness) and confirmed P. falciparum infection.
Sampling Method: Non-Probability Sample
Enrollment: 399 (Actual)
Dates: Start 2016-09-16 (Actual); Primary Completion 2018-09-06 (Actual); Study Completion 2018-09-06 (Actual)

PRIMARY OUTCOMES:
Percent prevalence of kelch13 mutants (marker of resistance to artemisinins) | 2 years

SECONDARY OUTCOMES:
Percent prevalence of specimens with pfmdr1 copy number >1 (marker of resistance to mefloquine) | 2 years
Visualization and dissemination of molecular marker prevalence data to inform public health officials, researchers, policymakers and key stakeholders | 2 yeas

CONTACTS AND LOCATIONS:
Locations (1):
- Study clinic, Komé, Doba, Chad

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Das S, Kerah-Hinzoumbe C, Kebfene M, Srisutham S, Nagorngar TY, Saralamba N, Vongpromek R, Khomvarn T, Sibley CH, Guerin PJ, Imwong M, Dhorda M. Molecular surveillance for operationally relevant genetic polymorphisms in Plasmodium falciparum in Southern Chad, 2016-2017. Malar J. 2022 Mar 12;21(1):83. doi: 10.1186/s12936-022-04095-9. PMID 35279140